CLINICAL TRIAL: NCT03433365
Title: Lenalidomide Maintenance in Multiple Myeloma Patients Achieving at Least VGPR After Induction Therapy: Minimal Residual Disease Monitoring
Brief Title: Monitoring of Deep of Response During Lenalidomide Maintenance in MM Patients Achieving at Least Very Good Partial Response (MRD)
Acronym: MRD
Status: Completed | Type: Observational
Sponsor: Fondazione EMN Italy Onlus (Other)
Responsible Party: Sponsor
Other Study IDs: RV-MM-PI-0694
Record Dates: First submitted 2018-02-08; First posted 2018-02-14 (Actual); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — MRD determination will be performed using the tumor specific IgH rearrangement through allele specific real time PCR (ASO PCR). This technique is sensitive enough to detect one myeloma cells out of 105-106 normal cells and allows to perform quantitative evaluation too. This method for molecular MRD determination has already been published and in our laboratory has already been used for MRD analysis in MM. 2720 Thermal cyclers (Applied Biosystems, Carlsbad, California, USA) and the AbiPrism 7900HT (Applied Biosystems, Carlsbad, California, USA) will be employed to analyze MRD using qualitative and quantitative PCR approach. Both nested qualitative and real time quantitative PCR will be employed in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Potential study subjects will sign an informed consent prior undergoing any study related procedure. Patients enrolled in this study will receive Lenalidomide-based regimen as maintenance therapy according to their previous decided therapeutic schedule. All consecutive patients treated with Lenalidomide-based regimen as maintenance therapy and with inclusion criteria will be asked to participate to this study.
  Interventions: Other: MRD analysis

INTERVENTIONS:
Other: MRD analysis — To collect 2 samples for MRD analysis in patients treated with Lenalidomide
  Other Names: No intervention_Observational study

SUMMARY:
This is an italian multicenter study to determine whether maintenance treatment with Lenalidomide-based regimen significantly increases the rate of molecular remission in patients achieving at least a VGPR after therapy with new drugs combination. No changing in the planned therapy will be made according to MRD results. A total of 70 patients with newly diagnosed MM who are 18 years of age or older and who meet all of the eligibility criteria may be enrolled in this study.

Potential study subjects will sign an informed consent prior undergoing any study related procedure. Patients enrolled in this study will receive Lenalidomide-based regimen as maintenance therapy according to their previous decided therapeutic schedule. All consecutive patients treated with Lenalidomide-based regimen as maintenance therapy and with inclusion criteria will be asked to participate to this study.

No additional drugs will be administrated for this study whose aim is to monitor the MRD on bone marrow aspirate and peripheral blood of patients during maintenance therapy with Lenalidomide-based regimen.

DETAILED DESCRIPTION:
Patients entering the study will signed an informed consent and will undergo bone marrow aspiration and peripheral blood examination. On both these two tissues the MRD analysis reaching for myeloma cells.

During the treatment period, all patients will attend study center visits every 4 weeks, until development of confirmed Progressive Disease (PD). During this visits the patients will undergo physical evaluation and routine blood control will be performed to monitor response to therapy and side effects.

When a patient develops a PD requiring the beginning of a new treatment, the patient interrupts the MRD monitoring but will be followed for survival every 2 months via telephone or office visit.

ELIGIBILITY:
Inclusion Criteria:

* Patient is, in the investigator(s) opinion, willing and able to comply with the protocol requirements.
* Patient has given voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to their future medical care.
* Patient has achieved at least a Very Good Partial Response (VGPR) before starting maintenance therapy
* Availability of a bone marrow sample at diagnosis stored in the Institution tissue bank to create patient-specific probes derived from IgH rearrangement
* Patients must receive Lenalidomide-based regimen as maintenance after a first line therapeutic approach
* Patient is 18 years old at the time of signing the informed consent
* Patient has a Karnofsky performance status ≥ 60%.
* Patient has a life-expectancy > 6 months
* Patient has HBV, HCV and HIV negative test.
* Patients must have normal ECG and NYHA ≤ 2; an evaluation of ejection fraction by ECHO or MUGA is optional
* Patients must be informed on acute and late toxicity of Lenalidomide treatment and must sign an informed consent.

Exclusion Criteria:

* Any serious medical condition, including the presence of laboratory abnormalities, which places the subject at an unacceptable risk if he or she participates in this study or confounds the experimental ability to interpret data from the study.
* Achieving of a PR or less before starting maintenance therapy
* Pregnant or lactating women. A serum β-hCG pregnancy test must be performed at the Screening visit, for female patients of child-bearing potential. If the test is positive, the patient must be excluded from the study. Confirmation that the patient is not pregnant must be established by a negative serum or urinary pregnancy test with the result obtained 1 day prior to the Baseline visit (or the day of the visit if results are available before drug delivery). A pregnancy test is not required for naturally post-menopausal women (who have not had menses at any time in the preceding 24 consecutive months) or surgically sterilised women (hysterectomy, bilateral ovariectomy, bilateral salpingectomy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential study subjects will sign an informed consent prior undergoing any study related procedure. Patients enrolled in this study will receive Lenalidomide-based regimen as maintenance therapy according to their previous decided therapeutic schedule.
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
MRD conversion | 2 years
  Rate of conversion from MRD positive to MRD negative during maintenance therapy (qualitative PCR approach)
Tumour load | 2 years
  Rate of patients with a reducing or increasing tumour load during therapy (quantitative real time PCR approach)
Molecular relapse | 2 years
  Rate of molecular relapse

SECONDARY OUTCOMES:
MRD negativity | 2 years
  MRD negativity duration during lenalidomide maintenance treatment
Molecular relapse | 2 years
  Time from diagnosis to molecular relapse. Evaluate if molecular relapse can be considered an early biomarker of relapse
Peripheral blood compared with bone marrow | 2 years
  Evaluate MRD negativity on peripheral blood samples and compare it with MRD analysis conducted on bone marrow samples
Overall Survival | 2 years
  Time from diagnosis to death in patients who achieved a molecular remission. Compare these results with the overall population

CONTACTS AND LOCATIONS:
Locations (1):
- AOU Città della Salute e della Scienza di Torino, Torino, Italy

IPD SHARING:
Plan to Share IPD: No